CLINICAL TRIAL: NCT07182357
Title: ENGAGE-D: Designing Care Management for Hospice Transitions for Persons Living With Advanced Dementia
Brief Title: Designing Care Management for Hospice Transitions for Persons Living With Advanced Dementia
Acronym: ENGAGE-D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Visiting Nurse Service of New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: i24-00426
Record Dates: First submitted 2025-06-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease and Related Dementias
Keywords: hospice care; care transitions; Alzheimer's disease and related dementias
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a Stage 1b clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia Care Management Checklist for Hospice Transitions (Experimental): The care management checklist will be administered to care partners by care managers during an outreach call to discuss the person with dementia's care and clinical needs. In this conversation, they will use the checklist to ask questions regarding care needs, decision-making considerations (healthcare proxy, etc), end-of-life dementia education, social and cultural needs, and potential care transitions.
  Interventions: Behavioral: Dementia Care Management Checklist for Hospice Transitions

INTERVENTIONS:
Behavioral: Dementia Care Management Checklist for Hospice Transitions — Intervention: After appropriate care partners of hospice-eligible PLWD are identified who will be receiving the checklist intervention, care managers will perform telephonic outreach to engage them in a conversation about care needs (as they would in typical clinical practice). The telephonic outreach will be followed up with a recommendation for follow up by a medical provider who may conduct a hospice care assessment and engage the care partner in decision-making surrounding the hospice referral and enrollment process.
  This intervention was co-designed with care partners, home healthcare professionals, administrators, and medical providers. It is meant to be comprehensive and speak to the needs of all relevant parties engaged in the care of persons with dementia. It is developed so that it can be scaled and implemented widely.

SUMMARY:
This study will test a care management intervention to guide end-of-life care and hospice transitions for persons with dementia and their care partners receiving home healthcare and ascertain feasibility, acceptability, fidelity, and usability of a dementia care management hospice transitions checklist. This study will also examine hospice enrollment, time to enrollment, and care partner satisfaction with the intervention. The intervention will be delivered within usual care management within a large home healthcare agency.

DETAILED DESCRIPTION:
This study has the following design: Unblinded, Non-Randomized, Single-Arm Intervention Study (Feasibility Trial). In this study, the team will pilot test the care management checklist intervention with care partners of persons with dementia. This intervention will be tested for feasibility (primary outcome), acceptability, fidelity, and usability (secondary) for in a single arm feasibility trial. The intervention will be administered (NIH Stage 1B) within usual care management for hospice transitions with care partners of PLWD. This study will also examine hospice enrollment and time to enrollment, and care partner satisfaction with the intervention.

The study population includes care partners and persons living with dementia; HHC professionals who engage in hospice transitions care management with care partners of PLWD (e.g., care managers who are nurses or social workers) and field nurses; Medical providers who engage in hospice transitions communication (e.g., home care physicians and nurse practitioners); HHC administrators who oversee and manage the delivery of care management prior to hospice transitions.

ELIGIBILITY:
Inclusion:

Care Partners and PLWD Dyad:

1. Care partners of PLWD who have a diagnosis of moderate to severe dementia.
2. Able to provide informed consent

HHC Professionals:

Care Managers and Field Nurses:

1. Care managers who regularly engage hospice transitions with care partners of PLWD
2. Age 18 or older

Medical Providers:

1. Medical providers (e.g., physicians and nurse practitioners) who refer patients for hospice enrollment.
2. Age 18 or older

HHC Administrators:

1. Home healthcare administrators who work with the Certified Home Health Agency or the Advanced Illness Management Program that refers patients to hospice care
2. Age 18 or older

Exclusion

Care Partner and PLWD Dyad

1. Under age 18
2. Care partners who are caring for PLWD with Mild Cognitive Impairment
3. PLWD with Mild Cognitive Impairment

HHC Professionals: Care Managers, Medical Providers, Administrators

1. Do not have experience managing hospice transitions for PLWD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Dementia Care Management Hospice Transitions Checklist | After enrollment and study participation, we will collect feasibility data within 1 month after intervention receipt.
  The primary outcome is feasibility. Feasibility will be measured for each group including recruitment and retention rates, rate of completion of the intervention as the proportion of individuals who use and receive the intervention, and whether the different components of the intervention are achievable.

SECONDARY OUTCOMES:
Acceptability of the Dementia Care Management Hospice Transitions Checklist | After intervention delivery, we will collect secondary outcome data within 1 month.
  The secondary outcome is acceptability. Acceptability will be reflected in process measures required in a transitional care management intervention. For example, intervention components will be measured including if the care manager/interventionist successfully receives the training and resources to successfully deliver the intervention and the number of HHC professionals for whom the intervention was acceptable. Outcome measure: Percentage of participants who find the intervention acceptable.

OTHER OUTCOMES:
Fidelity | To be measured within 1 month of intervention delivery.
  Fidelity will be assessed through healthcare professional adherence to study protocols and consistency in delivery of the intervention over time. Fidelity will be measured by assessing frequency of adherence to study protocols and pre-specified data collection processes and procedures (through participant response questionnaire). The percentage of individuals who maintained fidelity will also be measured.
Usability | To be measured within 1 month of intervention delivery.
  Usability will also be assessed and measured based on the percentage of people for whom the intervention was successfully usable (care partners and HHC professionals) and whether the checklist training and integration into care management is practicable. Usability will be measured as yes/no binary responses in a follow up questionnaire.
Hospice Enrollment and Time to Enrollment | Hospice enrollment and time to enrollment (of the person with dementia) will be measured at 1 and 6 months after intervention receipt.
  We will assess hospice enrollment and time to enrollment of the person with dementia (using the electronic health record) after the intervention.
Care Partner Satisfaction | To be measured within 1 month of intervention receipt.
  Care partner satisfaction will be evaluated using the 20-item Family Satisfaction with Advanced Cancer Care (FAMCARE), which has been validated for use in dementia care.
  Scoring the Original 20-Item FAMCARE Scale Identify the Scale's Items: The scale consists of 20 individual items designed to assess various aspects of care.
  Apply Likert Scale Scoring: Each item is rated on a 5-point Likert scale, with responses typically including:
  Very Satisfied Satisfied Undecided Dissatisfied Very Dissatisfied
  Calculate the Overall Score: The overall score is the sum of the responses to all 20 items.
  Interpret the Score: A higher total score signifies greater satisfaction with the healthcare provided to the patient and themselves. If a family member rates their satisfaction on a 5-point scale from 1 (Very Dissatisfied) to 5 (Very Satisfied) for all 20 items, then a higher sum of these ratings (e.g., close to 100) would indicate high satisfaction, while a lower sum is lower satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Rory Meyers College of Nursing and VNS Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified and redacted focus group and/or interview transcripts and coding summaries may be shared. De-identified intervention outcome measurement data and care partner satisfaction data may be shared. Study protocols and analysis plans will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available as soon as possible or at the time of associated publication. All data to be shared will be shared by the close of the reward. Data will be made available, at minimum, for seven years.
Access Criteria: All dataset(s) that can be shared will be deposited in the National Institute on Aging (NIA) National Alzheimer's Coordinating Center (NACC).

REFERENCES:
- [Background] Murali KP, Carpenter JG, Kolanowski A, Bykovskyi AG. Comprehensive Dementia Care Models: State of the Science and Future Directions. Res Gerontol Nurs. 2025 Jan-Feb;18(1):7-16. doi: 10.3928/19404921-20241211-02. Epub 2025 Jan 1. PMID 39836766
- [Background] Murali KP, Gogineni S, Bullock K, McDonald M, Sadarangani T, Schulman-Green D, Brody AA. Interventions and Predictors of Transition to Hospice for People Living With Dementia: An Integrative Review. Gerontologist. 2025 Apr 9;65(5):gnaf046. doi: 10.1093/geront/gnaf046. PMID 39903194